CLINICAL TRIAL: NCT03237728
Title: Randomized, Double-blind Placebo-controlled Clinical Study to Assess Safety, Tolerance, Pharmacokinetics, Pharmacodynamic of Multiple-dose Kukoamine B Mesilate in Sepsis Patients
Brief Title: Study of Multiple-dose Kukoamine B Mesilate in Sepsis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Chasesun Pharmaceutical Co., LTD (Industry)
Collaborators: Southwest Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HR-KB104
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2019-04

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0.06mg/kg,KB and Placebo (Experimental): Group A:0.06mg/kg,Q8h,Day1-Day7
  Interventions: Drug: 0.06mg/kg,KB; Drug: Placebos
- 0.12mg/kg,KB (Experimental): Group B:0.12mg/kg,Q8h,Day1-Day7
  Interventions: Drug: 0.12mg/kg,KB
- 0.24mg/kg,KB (Experimental): Group C:0.24mg/kg,Q8h,Day1-Day7
  Interventions: Drug: 0.24mg/,KB
- Placebos (Experimental): Group D:Placebos,Q8h,Day1-Day7
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: 0.06mg/kg,KB — 0.06mg/kg,Q8h,Day1-Day7
  Arms: 0.06mg/kg,KB and Placebo
Drug: 0.12mg/kg,KB — 0.12mg/kg,Q8h,Day1-Day7
  Arms: 0.12mg/kg,KB
Drug: 0.24mg/,KB — 0.24mg/kg,Q8h,Day1-Day7
  Arms: 0.24mg/kg,KB
Drug: Placebos — Placebos,Q8h,Day1-Day7
  Arms: 0.06mg/kg,KB and Placebo; Placebos

SUMMARY:
Phase I study of multiple-dose Kukoamine B Mesilate in Sepsis Patients

DETAILED DESCRIPTION:
To Assess Safety, Tolerance, Pharmacokinetics, Pharmacodynamic of multiple-dose Kukoamine B Mesilate in Sepsis Patients

ELIGIBILITY:
Inclusion Criteria:

1. The age of ≥ 18 years of age and ≤ 70 years of age, gender is not limited;
2. Confirmed or suspected bacterial infection (refer to Appendix 5);
3. Infection-related organ failure does not exceed 24 hours; organ failure is defined as circulation, (SOFA) ≥ 3 points in at least one organ or system of the respiratory, kidney, liver, coagulation and central nervous system;
4. The time interval between the selection of the test drug and the test drug is not more than 8 hours;
5. Infertility test for women of childbearing age;
6. Childbearing age within six months without child care plan and agreed to take effective measures during the study of contraception;
7. Patients or legal representatives signed informed consent.

Exclusion Criteria:

1. Pregnant or lactating women, or unable to take effective measures of contraception;
2. Patients are expected to live less than 28 days due to basic diseases, such as poor control of malignant tumor, cardiac arrest in 30 days, and end-stage lung disease.
3. The patient has the following chronic organ dysfunction or immunosuppression (based on the chronic health scoring assessment of the APACHE II score) : a) heart: New York heart association cardiac function IV; B) breathing: chronic obstructive, obstructive, or vascular lung disease can lead to severe restrictions on activities, i.e. the inability to go upstairs or to do housework; Or clear chronic hypoxia, CO2 retention, secondary real erythrocyte, severe pulmonary hypertension (> 40 mmHg) or respiratory muscle dependence; C) kidneys: receiving long-term dialysis; D) liver: liver cirrhosis confirmed by biopsy and clear portal hypertension; The upper digestive tract hemorrhage caused by portal hypertension; Or previous liver failure/hepatic encephalopathy/hepatic coma; E) of immune function: accept the treatment of impact resistance to infection, such as immune suppression therapy, chemotherapy, radiation therapy, or for a long time the recent use of high doses of hormones), or sickness impact resistance to infection, such as leukemia, lymphoma and AIDS);
4. Solid organ or bone marrow transplantation;
5. Plant survival status;
6. The following conditions occurred within 4 weeks prior to infection: a) acute pulmonary embolism; B) transfusion response; C) acute coronary syndrome;
7. Confirmed or highly suspected of acute infectious diseases such as viral hepatitis activity and active tuberculosis;
8. Patients with sinus bradycardia (less than 60 per minute);
9. Severe anemia (hemoglobin < 7.0 g/dL);
10. Uncontrolled bleeding in the past 24 hours;
11. Large area burns or chemical burns (III degree burns area > 30% BSA);
12. The average arterial pressure was < 65 mmHg after adequate liquid resuscitation and vasoactive drug therapy.
13. Acute myeloid hematopoiesis was characterized by a lack of severe granulocytes (ANC < 500 / mm3), or severe thrombocytopenia (< 20,000 / mm3);
14. Allergic to the active ingredient or its auxiliary materials;
15. The medication patients are using may severely affect the metabolism of the drug;
16. Patients and (or) legal representatives have signed an unresuscitation (DNR), or decided to withdraw life support (withdraw) or restrict life support for the intensity (of the patient) and sign the informed consent form;
17. Participated in clinical intervention test in 3 months;
18. The subject is a researcher or his immediate family member, or may have improper informed consent;
19. The attending physician considers it inappropriate for the patient to participate in this test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Day-1 to Day8
  AE, physical examination, monitoring of vital signs, Laboratory examination etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hu XY, Zhang W, Wang D, Sun Y, Hu Z, Zang B, Feng Y, Wang H, Zhou J, Zhao Q, Liu H, Wang T, Jiang W, Wang CY, Jin C, Dong K, Chen S, Yao X, Hu P, Du B; China Critical Care Clinical Trials Group (CCCCTG). Safety, tolerability, pharmacokinetics, and efficacy of kukoamine B in patients with sepsis: A randomized phase IIa trial. J Crit Care. 2023 Aug;76:154294. doi: 10.1016/j.jcrc.2023.154294. Epub 2023 Apr 26. PMID 37116228